CLINICAL TRIAL: NCT01288404
Title: A Pilot Study of Subconjunctival Bevacizumab Injection in Impending Recurrent Pterygium
Brief Title: Randomized Controlled Trial of Subconjunctival Bevacizumab Injection in Impending Recurrent Pterygium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Kaevalin Lekhanont, Ramathibodi Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 055217
Record Dates: First submitted 2011-02-01; First posted 2011-02-02 (Estimated); Last update posted 2011-02-02 (Estimated); Status verified 2011-01

CONDITIONS: Pterygium of the Conjunctiva and Cornea
Keywords: Bevacizumab, impending recurrent pterygium
MeSH Terms: conditions — Corneal Diseases | interventions — Fluorometholone; Bevacizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Placebo Comparator): topical 0.1% fluorometholone eye drops
  Interventions: Drug: Fluorometholone
- Bevacizumab group 1 (Active Comparator): Bevacizumab 1.25 mg/0.05mL
  Interventions: Drug: Bevacizumab
- Bevacizumab group 2 (Active Comparator): Bevacizumab 2.5 mg/0.1mL
  Interventions: Drug: Bevacizumab
- bevacizumab group 3 (Active Comparator): bevacizumab 3.75 mg/0.15mL
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Fluorometholone — topical 0.1% fluorometholone eye drops 4 times daily for 4 weeks
  Other Names: FML eye drops
  Arms: Control
Drug: Bevacizumab — subconjunctival bevacizumab 1.25 mg/0.05mL
  Other Names: Avastin
  Arms: Bevacizumab group 1
Drug: Bevacizumab — subconjunctival bevacizumab 2.5 mg/0.1mL
  Other Names: Avastin
  Arms: Bevacizumab group 2
Drug: Bevacizumab — subconjunctival bevacizumab 3.75 mg/0.15mL
  Other Names: Avastin
  Arms: bevacizumab group 3

SUMMARY:
Hypothesis: Subconjunctival bevacizumab injection may potentially suppress neovascularization in pterygium, preventing or retarding the progression of recurrence.

DETAILED DESCRIPTION:
1. Impending recurrent pterygium
2. Anti-VEGF therapy

   * Bevacizumab
   * Subconjunctival injection
   * Suppress neovascularization

ELIGIBILITY:
Inclusion Criteria:

1. Impending recurrent pterygium developed within 6 months following pterygium surgery either simple excision or excision with grafting.
2. Failure of conventional topical anti-inflammatory therapy for impending recurrent pterygium which was defined by the progression of fibrovascular tissue over the excised area despite receiving treatment.
3. No history of any adjunctive treatment such as MMC, 5-FU, periocular injection of corticosteroids and beta radiation.
4. No other ocular surface pathologies or coexisting ocular diseases.
5. No other ocular surgeries within the previous 6 months.
6. No history of allergy to the medications used in this study.
7. Good compliance with the study regimen and availability for the duration of the entire study period.

Exclusion Criteria:

1. Platelet disorders
2. Hypertension
3. Pregnant or lactating women

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-01; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Severity of impending recurrent pterygium | 3 months

SECONDARY OUTCOMES:
Visual analog scales | 3 months
Adverse reactions | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kaevalin Lekhanont, MD, Principal Investigator — Ramathibodi Hospital
Locations (1):
- Ramathibodi Hospital, Bangkok, Bangkok, Thailand